CLINICAL TRIAL: NCT05527431
Title: High Flow Nasal Cannula vs Noninvasive Ventilation in Patients With Hypoxic Respiratory Failure Following Blunt Chest Trauma, a Randomized Clinical Trial
Brief Title: High Flow Nasal Cannula vs Noninvasive Ventilation in Patients With Hypoxic Respiratory Failure Following Blunt Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAMSU R 115/ 2022
Record Dates: First submitted 2022-08-18; First posted 2022-09-02 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-08

CONDITIONS: Blunt Injury of Thorax
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high flow nasal cannula (Active Comparator)
  Interventions: Device: high flow nasal cannula
- noninvasive mechanical ventilation (Active Comparator)
  Interventions: Device: noninvasive ventilation

INTERVENTIONS:
Device: high flow nasal cannula — high flow nasal cannula
  Arms: high flow nasal cannula
Device: noninvasive ventilation — noninvasive ventilation
  Arms: noninvasive mechanical ventilation

SUMMARY:
to compare high flow nasal cannula against noninvasive ventilation in patients with non-sever blunt chest trauma in improvement of oxygenation, need for intubation and mechanical ventilation within 28 days

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 y,
* Willing and able to provide written informed consent prior to performing study procedures,
* currently hospitalized and requiring medical care for non-sever blunt chest trauma (abbreviated injury severity scale ≤ 2) SpO2 90% or less while breathing 10 L/min.

Exclusion Criteria:

* Contraindications of noninvasive ventilation (face trauma or surgery, airway obstruction, upper gastrointestinal tract bleeding, disturbed level of consciousness), -smoker
* intubation for any cause other than respiratory cause

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | 3 successive days
  mean value of three successive PaO2/FiO2 ratio in mmHg between both groups

SECONDARY OUTCOMES:
Discomfort score | 3 successive days
  Discomfort related to oxygen delivery devices will be evaluated using a 10- point numeric scale which low number is low discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No